CLINICAL TRIAL: NCT05936203
Title: Management of Prolonged Aerobic Exercise in Patients With Type 1 Diabetes on Advanced Technologies
Acronym: MARTA-walk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Annuzzi, Professor, Medical Doctor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Prot. 14/22
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Type1diabetes
Keywords: prolonged aerobic exercise; hybrid artificial pancreas; carbohydrates supplementation; insulin therapy

STUDY DESIGN:
Intervention Model Description: Randomized crossover clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Target (Experimental): Setting a higher glucose target starting from 1 hour before until the end of walk.
  Interventions: Other: Insulin therapy adjustment
- Snack (Experimental): Consumption of 15 g of complex carbohydrates as whole grain crackers every 30 minutes, during the 4 hours of walk.
  Interventions: Other: Nutritional adjustment
- Target + Snack (Experimental): Combination of both Target and Snack interventions.
  Interventions: Other: Combination of strategies

INTERVENTIONS:
Other: Insulin therapy adjustment — Strategies used to manage glucose control during a prolonged aerobic exercise
  Arms: Target
Other: Nutritional adjustment — Strategies used to manage glucose control during a prolonged aerobic exercise
  Arms: Snack
Other: Combination of strategies — Strategies used to manage glucose control during a prolonged aerobic exercise
  Arms: Target + Snack

SUMMARY:
The purpose of this study is to compare three different therapeutic and nutritional approaches during a prolonged aerobic exercise in moderately active type 1 diabetes people using advanced technologies, to identify the best strategy for the management of this type of exercise. Participants will be randomly assigned to different interventions in three different occasions: insulin therapy adjustment; nutritional adjustment; combination of insulin and nutritional adjustment.

DETAILED DESCRIPTION:
Regular exercise is recommended in people with type 1 diabetes (T1D) for its several health benefits (increased cardiovascular fitness, greater muscle strength, improved insulin sensitivity). However, therapeutic, and nutritional management of physical exercise is complex due to the multiple intra- and interindividual factors influencing glycemic response to exercise in T1D people. Glucose levels can increase, stay stable, or decrease depending on the type, duration, and intensity of exercise. During prolonged aerobic exercise, there is an increase in the risk of hypoglycemia also in patients using advanced technologies such as the hybrid artificial pancreas (HAP). The HAP consists of a continuous glucose monitoring (CGM) sensor and an insulin pump connected by a control algorithm that infuses insulin based on the glucose value recorded by the CGM sensor. With HAP there is the possibility to set a higher glucose target to make the insulin doses less aggressive during a scheduled session of physical exercise thus reducing the risk of hypoglycemia. However, there are different approaches, including insulin therapy adjustments or consumption of carbohydrates, proposed to minimize glycemic excursions during prolonged aerobic exercise in patients with T1D. Currently, the best strategy to manage physical exercise in people with type 1 diabetes on HAP, is not defined.

So, the aim of this study is to identify the optimal strategy for the management of prolonged aerobic exercise in moderately active T1D patients using hybrid artificial pancreas treatment. The exercise consists of an outdoor walk of 10 km over 4 hours and a height difference of 200-300 m. Each participant will be randomly assigned to three different therapeutic and nutritional interventions on three different occasions: 1)Target, which consists in setting a higher glucose target from 1 hour before until the end of the walk; 2) Snack, which consists of the consumption of 15 g of complex carbohydrates as whole grain crackers every 30 minutes, during the 4 hours of the walk; 3) Target+Snack consists in the combination of both Target and Snack interventions. Glycemic control expressed as CGM metrics and insulin doses delivered by HAP during the 4 hours of walks will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Using of hybrid artificial pancreas

Exclusion Criteria:

* Health conditions that may affect the safe performance of physical activity
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Time in Range | During 4 hours of walks in 3 different occasions
  Glucose concentrations at 5-min intervals will be downloaded from dedicated platforms and the percentage of time with a glycemia between 70-180 mg/dl during 4 hours of walks will be derived.
Insulin doses delivered | During 4 hours of walks in 3 different occasions
  Total insulin doses delivered by HAP during 4 hours of walks will be downloaded from the dedicated platforms.

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University Hospital, Naples, Italy